CLINICAL TRIAL: NCT00273793
Title: Increasing Contingency Management Success Using Shaping
Brief Title: Increasing Contingency Management Success in Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 045-0013-195; R01DA013304 (NIH)
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Results first posted 2012-06-07 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

ARMS (6):
- 1 (Experimental): Shaping intervention for hard-to-treat smokers
  Interventions: Behavioral: Contingency Management
- 2 (Active Comparator): fixed criterion intervention for hard-to-treat smokers
  Interventions: Behavioral: Contingency Management
- 3 (Other): Non contingent incentives available to hard to treat smokers
  Interventions: Behavioral: Contingency Management
- 4 (Experimental): Ascending incentives values used in Smokers with Early Success
  Interventions: Behavioral: Contingency Management
- 5 (Active Comparator): fixed value incentives are used in Smokers with Early Success
  Interventions: Behavioral: Contingency Management
- 6 (Other): Non contingent incentives are available to Smokers with Early Success
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — incentives are available for reduced smoking on each study visit which occur each weekday.

SUMMARY:
Incentives can be used to facilitate the acquisition of many healthy behaviors, such as smoking cessation. However, there is much room for improvement in the use of incentives. This study investigates how two aspects of providing incentives influence the effectiveness of using incentives to promote smoking cessation. One aspect is the criterion for providing incentives, e.g., whether to require smoking cessation before providing an incentive or to provide incentives following smoking reductions. The other aspect being investigated is whether it is best to use a fixed incentive amount or an amount that increases with continued cessation success.

ELIGIBILITY:
Inclusion Criteria: Daily Smokers smoking a pack or more of cigarettes a day who are able to report to the study site each work day for about 5 minutes for around 3 months. Subjects must also have a breath CO level indicative of smoking at this level, and most report smoking for at least two years. Subjects must intend on quitting smoking.

-

Exclusion Criteria: Participation in another study by this group within the past year. Inability to give informed consent. Incapable of attendance each workday during the morning hours.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2005-06; Primary Completion 2010-06 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Lamb, Ph.D., Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Smoking Cessation Laboratory, Department of Psychiatry, UTHSCSA, 7703 Floyd Curl Drive, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals smoking at least 15 cigarettes per day that are at least 18 years old, and deliver a breath CO level greater than or equal to 15 ppm were recruited in a University setting from the general community.
Pre-assignment Details: Five weekdaily visits that took about 5 minutes occurred before randomization. 328 individuals consented and of these 239 completed baseline and were randomized. Which set of three study arms individuals were randomly assigned to depended on whether they successfully delivered a C) < 3 ppm during this baseline for which they earned an incentive.
Groups:
- Shaping Intervention for Hard-to-treat Smokers: Shaping intervention for hard-to-treat smokers: Smokers who did not deliver a breath CO < 3 ppm in first five weekday sessions randomly assigned to receive incentives based upon a percentile schedule.
- Fixed Criterion Intervention for Hard-to-treat Smokers: fixed criterion intervention for hard-to-treat smokers: Smokers who did not deliver a breath CO < 3 ppm in first five weekday sessions randomly assigned to receive incentives for COs < 3 ppm.
- Non Contingent Incentives Available to Hard to Treat Smokers: Non contingent incentives available to hard to treat smokers: Smokers who did not deliver a breath CO < 3 ppm in first five weekday sessions randomly assigned to receive incentives non-contingently on a random basis.
- Ascending Incentives Values Used in Smokers With Early Success: Ascending incentives values used in Smokers with Early Success: Smokers who did deliver a breath CO < 3 ppm in first five weekday sessions randomly assigned to receive incentives that escalate in value with each delivery.
- Fixed Value Incentives Are Used in Smokers With Early Success: fixed value incentives are used in Smokers with Early Success: Smokers who did deliver a breath CO < 3 ppm in first five weekday sessions randomly assigned to receive incentives that are fixed in value
- Non Contingent Incentives Are Available to Smokers With Early: Non contingent incentives are available to Smokers with Early Success: Smokers who did deliver a breath CO < 3 ppm in first five weekday sessions randomly assigned to receive incentives that are non-contingently delivered on a random basis.
Period: Overall Study
Arm/Group | Shaping Intervention for Hard-to-treat Smokers | Fixed Criterion Intervention for Hard-to-treat Smokers | Non Contingent Incentives Available to Hard to Treat Smokers | Ascending Incentives Values Used in Smokers With Early Success | Fixed Value Incentives Are Used in Smokers With Early Success | Non Contingent Incentives Are Available to Smokers With Early
Started | 36 | 38 | 18 | 60 | 58 | 29
Completed | 36 | 38 | 18 | 60 | 58 | 29
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shaping Intervention for Hard-to-treat Smokers | Fixed Criterion Intervention for Hard-to-treat Smokers | Non Contingent Incentives Available to Hard to Treat Smokers | Ascending Incentives Values Used in Smokers With Early Success | Fixed Value Incentives Are Used in Smokers With Early Success | Non Contingent Incentives Are Available to Smokers With Early | Total
Number analyzed (Participants) | 36 | 38 | 18 | 60 | 58 | 29 | 239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 37 | 18 | 59 | 58 | 29 | 237
  >=65 years | 0 | 1 | 0 | 1 | 0 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 44.8 (12.2) | 43.3 (12.8) | 43.1 (11.2) | 41.9 (12.9) | 41.3 (11.8) | 40.6 (10.0) | 42.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 7 | 25 | 26 | 16 | 98
  Male | 24 | 26 | 11 | 35 | 32 | 13 | 141
Region of Enrollment [Number; unit: participants]
  United States | 36 | 38 | 18 | 60 | 58 | 29 | 239

OUTCOME MEASURES:

1. Primary Outcome: Breath Carbon Monoxide Levels Indicating Smoking Abstinence During the Study, i.e., the Number of Breath Samples With Carbon Monoxide (CO) Levels Less Than 3 Parts Per Million (Ppm)
Time Frame: daily for breath CO
Population: all subjects randomized to condition
Measure: Median (Inter-Quartile Range); unit: number breath samples < 3 ppm CO
Arm/Group | Shaping Intervention for Hard-to-Treat Smokers | Fixed Criterion Intervention for Hard-to-Treat Smokers | Non Contingent Incentives Available to Hard-to-Treat Smokers | Ascending Incentive Values Used in Smokers With Early Success | Fixed Value Incentives Are Used in Smokers With Early Success | Non Contingent Incentives Are Available to Smokers With Early
Number analyzed (Participants) | 36 | 38 | 18 | 60 | 58 | 29
number breath samples < 3 ppm CO | 2 [0 to 12.5] | 3.5 [0 to 39] | 0 [0 to 12.0] | 58.5 [15 to 64] | 49.5 [25 to 61] | 28 [6 to 59]

2. Secondary Outcome: Average Number Cigarettes Reported Smoked Each Day in the Past Week Measured at Follow-up Six Months After Entry Into the Study
Description: average number cigarettes reported smoked each day in the past week at follow up six months after study entry
Time Frame: past week at follow-up six months after study entry
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Shaping Intervention for Hard-to-Treat Smokers | Fixed Criterion Intervention for Hard-to-Treat Smokers | Non Contingent Incentives Available to Hard-to-Treat Smokers | Ascending Incentive Values Used in Smokers With Early Success | Fixed Value Incentives Are Used in Smokers With Early Success | Non Contingent Incentives Are Available to Smokers With Early
Number analyzed (Participants) | 34 | 28 | 14 | 41 | 43 | 23
cigarettes per day | 12.8 (12.0) | 12.6 (7.7) | 15.1 (8.2) | 11.5 (9.9) | 11.1 (8.2) | 8.2 (7.2)

ADVERSE EVENTS:
Arm/Group | Shaping Intervention for Hard-to-treat Smokers | Fixed Criterion Intervention for Hard-to-treat Smokers | Non Contingent Incentives Available to Hard to Treat Smokers | Ascending Incentives Values Used in Smokers With Early Success | Fixed Value Incentives Are Used in Smokers With Early Success | Non Contingent Incentives Are Available to Smokers With Early
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/38 | 0/18 | 0/60 | 0/58 | 0/29
Other Adverse Events (participants affected / at risk) | 0/36 | 0/38 | 0/18 | 0/60 | 0/58 | 0/29

LIMITATIONS AND CAVEATS:
The study was conducted largely as planned. However the study was not designed to adequately test post-treatment outcomes, as this would not be justifiable unless during treatment differences were observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes